CLINICAL TRIAL: NCT00056459
Title: A Randomized, Double-blind, Placebo-controlled, Phase Lll Study in Patients With Metastatic Adenocarcinoma of the Colon or Rectum Who Are Receiving First-line Chemotherapy With Oxaliplatin/5-fluorouracil/Leucovorin With PTK787/ZK 222584 or Placebo
Brief Title: Study of Oxaliplatin/5-FU/Leucovorin Plus Vatalanib Versus Oxaliplatin/5-FU/Leucovorin in Patients With Metastatic Colorectal Cancer.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Bayer (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CPTK787 0135/306241; CONFIRM 1
Record Dates: First submitted 2003-03-13; First posted 2003-03-14 (Estimated); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms
Keywords: Colorectal Cancer; PTK787; Vatalanib; VEGF inhibitor; Oxaliplatin; Angiogenesis; Rectal Cancer; Colon Cancer; Colorectal Carcinoma; Colorectal Tumor
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — vatalanib

ARMS (2):
- 1 (Experimental): Oxaliplatin/5-FU/LV and PTK787/ZK 222584
  Interventions: Drug: Vatalanib
- 2 (Placebo Comparator): Oxaliplatin/5-FU/LV and placebo
  Interventions: Drug: Vatalanib

INTERVENTIONS:
Drug: Vatalanib
  Other Names: PTK787/ZK 222584

SUMMARY:
To compare treatment with oxaliplatin/5-FU/leucovorin plus vatalanib versus oxaliplatin/5-FU/leucovorin plus placebo in patients with colorectal cancer that has spread to other organs and are seeking first chemotherapy treatment

ELIGIBILITY:
Inclusion criteria:

* Patients with metastatic colorectal cancer coming for initial chemotherapy
* Documented metastatic colorectal cancer
* WHO Performance Status of 0, 1, or 2
* Measurable tumors
* Adequate hematologic status, liver and kidney function
* Life expectancy greater than 12 weeks
* Written informed consent obtained

Exclusion criteria:

* History or presence of central nervous system disease
* Patients with a history of another primary cancer within 5 years
* Prior chemotherapy for metastatic colorectal cancer
* Prior full field radiotherapy within 4 weeks or limited field radiotherapy within 2 weeks before entry to study
* Major surgery within 4 weeks or minor surgery within 2 weeks before entry to study
* Investigational drugs within 4 weeks before entry to study
* Prior therapy with anti-VEGF agents
* Any prior therapy with oxaliplatin or allergy to platinum-containing drugs
* Peripheral neuropathy with functional impairment
* Female patients who are pregnant or breast feeding
* Any severe or uncontrolled medical conditions which could prevent participation in study
* Patients who are taking Coumadin

Other protocol-defined inclusion / exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1168 (Actual)
Dates: Start 2003-02; Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Progression free survival | Throughout duration of study

SECONDARY OUTCOMES:
Time to progression | Throughout duration of study
Time to treatment failure | Throughout duration of study
Best overall response rate | Throughout duration of study
Tolerability and safety profile | Throughout duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Novartis / Schering AG, Germany, Study Chair — Novartis / Schering AG, Germany
Locations (211):
- United States (144):
  - Alabama Hematology/Oncology, Birmingham, Alabama
  - Palo Verde Hematology & Oncology, Glendale, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - Northeast Arkansas Clinic, Jonesboro, Arkansas
  - Highlands Oncology Group, Springdale, Arkansas
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - Providence St. Joseph Medical Center, Burbank, California
  - Compassionate Cancer Care Medical Group, Inc, Fountain Valley, California
  - California Oncology of the Central Valley, Fresno, California
  - Virginia K. Crosson Cancer Center, Fullerton, California
  - Ronald Yanagiharaa, M.D., Gilroy, California
  - Glendale Adventist Medical Center Cancer Center, Glendale, California
  - Pacific Shores Medical Group, Long Beach, California
  - Cancer Institute Medical Group, Los Angeles, California
  - USC/Norris Comprehensive Cancer Care Center, Los Angeles, California
  - Synergy Hematology-Oncology Medical Associates, Los Angeles, California
  - UCLA School of Medicine, Los Angeles, California
  - Eddie Hong-Lung Hu, M.D., Monterey Park, California
  - North Valley Hematology/Oncology Medical Group, Northridge, California
  - Ventura County Hematology-Oncology Specialists, Oxnard, California
  - Wilshire Oncology Medical Group, Pomona, California
  - Sierra View District Hospital, Porterville, California
  - The Lucy Curci Cancer Center, Rancho Mirage, California
  - Cancer Care Associates Medical Group, Inc., Redondo Beach, California
  - Pacific Hematology Oncology Associates, San Francisco, California
  - Santa Clara Valley Medical Center, San Jose, California
  - Sansum Santa Barbara Foundation Medical Clinic, Santa Barbara, California
  - Santa Barbara Hematology Oncology Medical Group, Inc., Santa Barbara, California
  - San Diego Cancer Center Medical Group, Vista, California
  - Colorado Cancer Research Program, Denver, Colorado
  - Jennifer Caskey, M.D., Wheat Ridge, Colorado
  - Davis, Posteraro and Wasser, MD's, LLP, Manchester, Connecticut
  - Connecticut Oncology Group, Middletown, Connecticut
  - Medical Oncology Hematology Consultants, Newark, Delaware
  - Washington Oncology-Hematology Center, Washington D.C., District of Columbia
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Boca Raton Comprehensive Cancer Center, Boca Raton, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - Memorial Healthcare System, Hollywood, Florida
  - Florida Oncology Associates, Jacksonville, Florida
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - Oncology Hematology Group of South Florida, Miami, Florida
  - Innovative Medical Research of South Florida, Miami Shores, Florida
  - Hematology Oncology Associates of Treasure, Port Saint Lucie, Florida
  - Florida Medical Clinic, PA, Zephyrhills, Florida
  - Peachtree Hematology and Oncology, Atlanta, Georgia
  - Coastal Hematology & Oncology, Savannah, Georgia
  - North Idaho Cancer Center, Coeur d'Alene, Idaho
  - Shelby D. Rifkin, M.D., Arlington Heights, Illinois
  - Monroe Medical Associates, Harvey, Illinois
  - Oncology Hematology Associates of Central Illinois, PC, Peoria, Illinois
  - Northshore Cancer Research Association, Skokie, Illinois
  - Midwest Cancer Research Group, Skokie, Illinois
  - Hematology-Oncology of Indiana, PC, Indianapolis, Indiana
  - Associated Physicians & Surgeons Clinic, L.L.C., Terre Haute, Indiana
  - Markey Clinical Oncology Research Program, Lexington, Kentucky
  - Norton Healthcare Pavilion, Louisville, Kentucky
  - Vijay Raghavan, M.D., Louisville, Kentucky
  - Louisiana Oncology Associates, Lafayette, Louisiana
  - LSU Medical Center, New Orleans, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - LSU Health Sciences Center, Shreveport, Louisiana
  - Maine Center for Cancer Medicine & Blood Disorders, Scarborough, Maine
  - St. Agnes Healthcare, Inc., Baltimore, Maryland
  - Kaiser Permanente, Rockville, Maryland
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - Josephine Ford Cancer Center, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Spectrum Health -- Cook Research Dept., Grand Rapids, Michigan
  - Hematology and Oncology Assoc. of Southern Mississippi, Jackson, Michigan
  - Oncology Care Associates, PLLC, Saint Joseph, Michigan
  - Providence Cancer Center, Southfield, Michigan
  - SMDC Health System, Duluth, Minnesota
  - Minnesota CGOP, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Metro Minnesota CCOP, Saint Louis Park, Minnesota
  - Heartland Hematology/Oncology Associates, Inc., Kansas City, Missouri
  - Kansas City Oncology and Hematology Group, Kansas City, Missouri
  - Missouri Cancer Care, PC, Saint Charles, Missouri
  - Saint Louis University, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Arch Medical Services Incorporated, St Louis, Missouri
  - North Central Montana Professional Building, Great Falls, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - The Methodist Cancer Center, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Nevada Cancer Center, Las Vegas, Nevada
  - The Center for Cancer and Hematologic Disease, Cherry Hill, New Jersey
  - St. Barnabas Cancer Center, Livingston, New Jersey
  - Hematology-Oncology Associates of New Jersey, Morristown, New Jersey
  - Southern Oncology and Hematology Associates, Vineland, New Jersey
  - Cooper Cancer Institute, Voorhees Township, New Jersey
  - New Mexico Cancer Care, Santa Fe, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - CR Wood Cancer Center, Glens Falls, New York
  - Cancer Research of Long Island, Great Neck, New York
  - Broome Oncology, Johnson City, New York
  - New York Oncology Hematology, Latham, New York
  - North Shore University Hospital, Manhasset, New York
  - Cancer Center at Nyack Hospital, Nyack, New York
  - Pluta Cancer Center, Rochester, New York
  - Carolina Medical Center, Charlotte, North Carolina
  - Mid-Dakota Clinic PC, Bismarck, North Dakota
  - Nashat Gabrail, M.D., Canton, Ohio
  - Mid Ohio Oncology/Hematology, Inc., Columbus, Ohio
  - Hematology Oncology Consultants, Inc., Columbus, Ohio
  - Meridia Cancer Institute, Mayfield Heights, Ohio
  - Cancer Care Associates, Oklahoma City, Oklahoma
  - Cancer Care Associates, Tulsa, Oklahoma
  - Kaiser Permanente Oncology Hematology, Portland, Oregon
  - Hershey Medical Center, Hershey, Pennsylvania
  - Monogahela Valley Hospital, Monongahela, Pennsylvania
  - University of Pennsylvania Abramson Cancer Center, Philadelphia, Pennsylvania
  - Allegheny Cancer Center, Pittsburgh, Pennsylvania
  - Charleston Hematology Oncology, Charleston, South Carolina
  - Charleston Cancer Center, Charleston, South Carolina
  - South Carolina Oncology Associates, Columbia, South Carolina
  - Cancer Center of the Carolinas, Greenville, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - The Jones Clinic, Germantown, Tennessee
  - Baptist Regional Cancer Center, Knoxville, Tennessee
  - University of Tennessee Cancer Institute, Memphis, Tennessee
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - Southwest Regional Cancer Center, Austin, Texas
  - Corpus Christi Cancer Center, Corpus Christi, Texas
  - Center for Oncology Research & Treatment, PA, Dallas, Texas
  - Oncology Consultants, Houston, Texas
  - H. Alejandro Preti, MD, PA, Houston, Texas
  - M.D. Anderson Cancer Center, Houston, Texas
  - Dr. Lee C. Drinkard, Irving, Texas
  - Scott & White Hospital, Temple, Texas
  - North Utah Associates, Ogden, Utah
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Southwestern Vermont Health Care, Bennington, Vermont
  - Danville Hematology and Oncology, Inc., Danville, Virginia
  - Northern Virginia Oncology Group, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Cancer Treatment Centers of America, Portsmouth, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - Western Washington Medical Group, Everett, Washington
  - Cascade Cancer Center, Kirkland, Washington
  - UW Health -- University of Wisconsin Comp, Madison, Wisconsin
  - Waukesha Memorial Hospital, Waukesha, Wisconsin
- Australia (5):
  - Adelaide
  - Garran
  - Nedlands
  - Wollongong
  - Woolloongabba
- Belgium (5):
  - Anderlecht
  - Antwerp
  - Brussels
  - Ghent
  - Wilrijk
- Brazil (4):
  - Porto Alegre
  - Porto Alegre RS
  - Salvador
  - São Paulo
- Canada (4):
  - Hamilton, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Toronto, Ontario
  - Sainte-Foy, Quebec
- Czechia (2):
  - Brno
  - Prague
- France (2):
  - Marseille
  - Strasbourg
- Germany (13):
  - Augsburg
  - Berlin
  - Cologne
  - Dessau
  - Erlangen
  - Eschweiler
  - Essen
  - Frankfurt
  - Hanover
  - Heidelberg
  - Kiel
  - Leipzig
  - Magdeburg
- Hungary (3):
  - Budapest
  - Győr
  - Szeged
- Italy (7):
  - Forlì
  - Genova
  - Milan
  - Modena
  - Roma
  - Rozzano
  - Torino
- GA Utrecht, Netherlands
- New Zealand (2):
  - Novartis Investigative Site, Hamilton
  - Palmerston North
- Coimbra, Portugal
- Slovakia (3):
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Žilina
- Spain (4):
  - Alicante
  - Madrid
  - Málaga
  - Zaragoza
- Stockholm, Sweden
- Switzerland (4):
  - Basel
  - Bern
  - Thun
  - Zurich
- Taiwan (3):
  - Tainan
  - Taipei
  - Taoyuan District
- United Kingdom (3):
  - Belfast
  - Leicester
  - Oxford

REFERENCES:
- [Derived] Hecht JR, Trarbach T, Hainsworth JD, Major P, Jager E, Wolff RA, Lloyd-Salvant K, Bodoky G, Pendergrass K, Berg W, Chen BL, Jalava T, Meinhardt G, Laurent D, Lebwohl D, Kerr D. Randomized, placebo-controlled, phase III study of first-line oxaliplatin-based chemotherapy plus PTK787/ZK 222584, an oral vascular endothelial growth factor receptor inhibitor, in patients with metastatic colorectal adenocarcinoma. J Clin Oncol. 2011 May 20;29(15):1997-2003. doi: 10.1200/JCO.2010.29.4496. Epub 2011 Apr 4. PMID 21464406